CLINICAL TRIAL: NCT02142192
Title: A Multicenter, Open-Label Immunogenicity and Safety Study of Subcutaneous Natalizumab 300 mg Administered to Subjects With Relapsing Multiple Sclerosis
Brief Title: Natalizumab Subcutaneous Immunogenicity and Safety Study
Acronym: SIMPLIFY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101MS207; 2014-000917-30 (EudraCT Number)
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- natalizumab (Experimental): natalizumab 300mg SC every 4 weeks for up to 12 treatment administrations (i.e. Day 1 through Week 44)
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the treatment arm
  Other Names: BG00002; Tysabri

SUMMARY:
The primary objective of this study is to evaluate the immunogenicity of natalizumab (BG00002) 300 mg subcutaneous (SC) administered to participants with relapsing multiple sclerosis (RMS). The secondary objectives of the study are to evaluate the safety of natalizumab SC injections and to evaluate the efficacy of natalizumab SC injections on relapses and on new magnetic resonance imaging (MRI) lesions.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have documented diagnosis of RMS at screening.
* Must fall within the therapeutic indications stated in the locally approved label for natalizumab.
* Must have an EDSS score from 0 to 6.5, inclusive.

Key Exclusion Criteria:

* Any prior use of natalizumab.
* Positive for anti-natalizumab antibodies at screening.
* Treatment with immunomodulatory injections (including IFN-β and glatiramer acetate) within 2 weeks prior to Screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2015-06-04 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with persistent anti-natalizumab antibodies | 48 weeks
  Persistent anti-natalizumab antibodies are defined as 2 positive anti-natalizumab test results separated by at least 6 weeks, with at least 1 positive test result occurring at or after the Week 24 Visit.

SECONDARY OUTCOMES:
Proportion of participants with transient anti-natalizumab antibodies | 48 weeks
Proportion of participants with post-injection adverse events (AEs) | 48 weeks
  Including hypersensitivity reactions, anaphylactic reactions and other AEs occurring within 1 hour after SC natalizumab dosing.
Proportion of participants with clinical relapse | 48 weeks
  This may include new or enlarging T2 lesion(s), as determined by magnetic resonance imaging (MRI). Clinical relapse is defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the neurologist.
Proportion of participants with gadolinium (Gd) enhancing lesion(s) as assessed by MRI. | 48 weeks
Proportion of Participants that experience Adverse Events and Serious Adverse Events | up to 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Liège

REFERENCES:
- See also: EudraCT Tabulated Result — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-000917-30/results